CLINICAL TRIAL: NCT04295642
Title: A 2-Part, Open Label, Adaptive, Single and/or Multiple Oral Dose, Safety, Tolerability, and Food Effect Trial of CVL-751 in Subjects With Parkinson's Disease
Brief Title: A 2-Part Trial of CVL-751 in Subjects With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-PD-005
Record Dates: First submitted 2020-01-24; First posted 2020-03-04 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Placebo Comparator): Will include 4 subjects (3 active + 1 placebo) that will receive a single 15mg dose with approximately 48 hours of confinement and a follow-up after 7 days.
  Interventions: Drug: CVL-751
- Part 2 (Experimental): 2A: will include 14 subjects to complete 12 with 28 days of dosing with 7 days (+/-2) of follow-up, with at least 14 days of confinement.
  -or- 2B: will include 20 subjects to complete 12 with 2 dosing days and 5 days of washout with 7 days (+/-2) of follow-up, with 4 days of confinement (may be increased up to 12 days at the investigators discretion).
  Interventions: Drug: CVL-751

INTERVENTIONS:
Drug: CVL-751 — Oral tablet

SUMMARY:
This trial will be a 2-part, adaptive, open label, single and/or multiple oral dose, safety, tolerability, food effect trial of CVL-751 in subjects with Parkinson's disease. Part 1 is a placebo-controlled, single dose cohort intended for assessment of safety and tolerability. In case of intolerable AEs, Part 2 would proceed as a multiple dose titration trial to achieve a 15 mg once daily dose while maintaining L-Dopa treatment (Part 2A). In case of a favorable tolerability profile in Part 1, Part 2B would proceed as a single dose trial (similar to Part 1), with discontinuation of L-Dopa for 24 hours (12 hours pre-Day 1 dose and 12 hours post-Day 1 dose).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 45 to 75 years, inclusive, at the time of signing the informed consent form (ICF).
2. Body mass index (BMI) of 17.5 to 38.0 kg/m2 and a total body weight >50 kg (110 lbs).
3. Subjects with a diagnosis of that is consistent with the UK Parkinson's Disease Society Brain Bank diagnostic criteria, with bradykinesia and motor asymmetry.
4. Must be modified Hoehn & Yahr (HY) Stage I - III inclusive.
5. Must be on a stable dose of L-Dopa of at least 300 mg daily in conjunction with a dopa-decarboxylase inhibitor (eg, L-Dopa/carbidopa or L-Dopa/benserazide) administered at least 3 times per day but no more than 6 times per day for at least 2 weeks prior to the Day 1 Visit. Must be willing and able to refrain from L-Dopa treatment (in Part 1 and Part 2B) as outlined in the schedule of assessments.
6. A female subject of childbearing potential (see Section 10.4, Appendix 4) who is sexually active with a nonsterilized male partner or male subject with a pregnant or a nonpregnant partner of childbearing potential must agree to use an acceptable or a highly effective method of contraception (see Section 10.4, Appendix 4) from signing of informed consent throughout the duration of the trial and for 7 days post last dose.
7. Capable of giving signed informed consent as described in Section 10.1.3 (Appendix 1), which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
8. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.
9. Capable of consuming the standard high-fat meal.

Exclusion Criteria:

1. Any significant Axis I psychiatric disease as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (American Psychiatric Association).
2. In the opinion of the investigator (or caregiver, as applicable), has signs/symptoms suggestive of clinically significant cognitive impairment that would interfere with the ability to comply with trial procedures.
3. Subjects with a Montreal Cognitive Assessment score <26.
4. History or clinical features consistent with an atypical parkinsonian syndrome (eg, ataxia, dystonia, clinically significant orthostatic hypotension).
5. Has a history of psychotic symptoms requiring treatment with an antipsychotic medication within the 12 months prior to signing ICF.
6. Subjects with epilepsy, or history of epilepsy, or conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), or who have increased risk of seizures as evidenced by history of electroencephalogram with epileptiform activity.

   Subjects with a history of febrile seizures only are allowed. Subjects with a history of head trauma with loss of consciousness requiring overnight hospitalization will be excluded as well.
7. Subjects with a current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological disease that, in the opinion of the investigator or medical monitor, could compromise either subject safety or the results of the trial.

   Medical conditions that are minor or well-controlled may be considered acceptable if the condition does not expose the subject to an undue risk of a significant AE or interfere with the assessments of safety or efficacy during the course of the trial. The medical monitor should be contacted in any instance where the investigator is uncertain regarding the stability of a subject's medical conditions(s) and the potential impact of the condition(s) on trial participation.
8. History of substance or alcohol-use disorder (excluding nicotine; Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria) within 2 years prior to signing the ICF.
9. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months prior to signing ICF.
10. If a current smoker, is unable to comply with the following guidelines: agrees not to smoke on the mornings of trial dosing days and for the entire trial dosing day until completion of all trial assessments for that day.
11. Subjects who answer "Yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 6 months OR Subjects who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Subjects who, in the opinion of the investigator, present a serious risk of suicide.
12. Subjects who have attempted suicide in the past.
13. Human immunodeficiency virus seropositive status or acquired immunodeficiency syndrome, acute or chronic hepatitis B or C, with HbsAg, or hepatitis C virus antibodies at screening.
14. Subjects with a positive drug screen for illicit drugs are excluded and may not be retested or rescreened. Subjects with a positive urine drug screen resulting from use of marijuana (any cannabinoids), prescription medications, over-the-counter medications, or products that, in the investigator's documented opinion, do not signal a clinical condition that would impact the safety of the subject or interpretation of the trial results may continue evaluation for the trial following consultation and approval by the medical monitor.
15. Subjects with a 12-lead electrocardiogram (ECG) demonstrating the following:

    • QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec.
16. Subjects with any of the following abnormalities in clinical laboratory tests at the Screening Visit, as assessed by the central laboratory and confirmed by a single repeat measurement, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 × upper limit of normal (ULN)
    * Total bilirubin ≥1.5 × ULN. Subjects with a history of Gilbert's syndrome may be eligible provided the direct bilirubin is <ULN.
17. Subjects with other abnormal laboratory test results, vital sign results, or ECG findings unless, based on the investigator's judgment, the findings are not medically significant and would not impact the safety of the subjects or the interpretation of the trial results. The medical monitor should be contacted to discuss individual cases, as needed.

    Tests with exclusionary results should be repeated to ensure reproducibility of the abnormality before excluding a subject based on criteria provided in the protocol. For ECGs, three consecutive recordings are required and if two of the three remain exclusionary, then the subject is not eligible for the trial.
18. Subjects taking other prohibited medication or who would be likely to require prohibited concomitant therapy during the trial (see Section 6.5).
19. Female subjects who are breastfeeding and/or who have a positive serum pregnancy test result prior to receiving IMP.
20. Any condition possibly affecting drug absorption (eg, gastrectomy).
21. Subjects with difficulty swallowing.
22. Subjects who are known to be allergic or hypersensitive to the IMP or any of its components.
23. Subjects who are known to be allergic or hypersensitive to contents of high-fat diet.
24. Subjects who have participated in any clinical trial within 60 days prior to signing the ICF or who participated in more than two clinical trials within the year prior to signing the ICF.
25. Any subject who, in the opinion of the sponsor, investigator, or medical monitor, should not participate in the trial.
26. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator.
27. Unwilling or unable to comply with the lifestyle modifications described in this protocol.
28. Subjects who participated in Part 1 of the trial are ineligible to participate in Part 2.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Single Dose: Peak Plasma Concentration | Day 1 to 12
  Peak Plasma Concentration (Cmax) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Single Dose:Area under the plasma concentration-time curve | Day 1 to 12
  Area under the plasma concentration-time curve (AUC) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Single Dose: Area under the plasma concentration-time curve from time zero to infinity | Day 1 to 12
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Single Dose: Time to Maximum Concentration | Day 1 to 12
  Time to Maximum Concentration (Tmax) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Multiple Dose: Peak Plasma Concentration | Day 16 to 29
  Peak Plasma Concentration (Cmax) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Multiple Dose: Area under the plasma concentration-time curve | Day 16 to 29
  Area under the plasma concentration-time curve (AUCτ) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions
Multiple Dose: Time to Maximum Concentration | Day 16 to 29
  Time to Maximum Concentration (Tmax) for CVL-751 and its metabolite (PF-06752844) under fasted and fed conditions

SECONDARY OUTCOMES:
Secondary Outcome (AE) Number of subjects with reported Treatment Emergent Adverse Events (TEAEs) | up to Day 35
  Number of subjects with reported Treatment Emergent Adverse Events (TEAEs)
Secondary Outcome (Labs) Number of subjects with clinically significant changes in laboratory measures | up to Day 35
  Number of subjects with clinically significant changes in laboratory measures
Secondary Outcome (ECGs)Number of subjects with Clinically significant changes in Electrocardiogram | up to Day 35
  Number of subjects with Clinically significant changes in Electrocardiogram measures (PR,RR,QT and QTcF)
Secondary Outcome (Vital Signs) Number of subjects with Clinically meaningful changes in Vital signs | up to Day 35
  Number of subjects with Clinically meaningful changes in Vital signs
Secondary Outcome (C-SSRS) - Change from baseline of the Columbia-Suicide Severity Rating Scale(C-SSRS) | up to Day 35
  Change from baseline of the Columbia-Suicide Severity Rating Scale(C-SSRS) The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, Study Director — Cerevel Therapeutics, LLC
Locations (2):
- United States (2):
  - CNS Network, Long Beach, California
  - Atlanta Center for Medical Research, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression, and mortality. 1967. Neurology. 2001 Nov;57(10 Suppl 3):S11-26. No abstract available. PMID 11775596
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Result] Nussbaum RL, Ellis CE. Alzheimer's disease and Parkinson's disease. N Engl J Med. 2003 Apr 3;348(14):1356-64. doi: 10.1056/NEJM2003ra020003. No abstract available. PMID 12672864
- [Result] Rascol O, Brooks DJ, Korczyn AD, De Deyn PP, Clarke CE, Lang AE. A five-year study of the incidence of dyskinesia in patients with early Parkinson's disease who were treated with ropinirole or levodopa. N Engl J Med. 2000 May 18;342(20):1484-91. doi: 10.1056/NEJM200005183422004. PMID 10816186
- [Result] Schrag A, Banks P. Time of loss of employment in Parkinson's disease. Mov Disord. 2006 Nov;21(11):1839-43. doi: 10.1002/mds.21030. PMID 16941456
- [Result] Yamamoto M, Schapira AH. Dopamine agonists in Parkinson's disease. Expert Rev Neurother. 2008 Apr;8(4):671-7. doi: 10.1586/14737175.8.4.671. PMID 18416667